CLINICAL TRIAL: NCT03365739
Title: Bioavailability and Pharmacokinetic Parameters of Mango Pulp Phytochemicals in Human Plasma
Brief Title: Bioavailability and Pharmacokinetics of Mango
Acronym: MG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: IRB#2017-064
Record Dates: First submitted 2017-11-13; First posted 2017-12-07 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Healthy Subjects
Keywords: Mango; Mango pulp phytochemicals bioavailability; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active Comparator 1 (Active Comparator): Treatment - Mango (pulp/flesh-500 g)
  Interventions: Dietary Supplement: Active Comparator 1
- Active Comparator 2 (Active Comparator): Mango (500 g) + Vitamin C (100 mg)
  Interventions: Dietary Supplement: Active Comparator 2
- Control Comparator (Placebo Comparator): Vitamin C (100 mg)
  Interventions: Dietary Supplement: Control Comparator

INTERVENTIONS:
Dietary Supplement: Active Comparator 1 — Mango (pulp/flesh) (500 g)
  Arms: Active Comparator 1
Dietary Supplement: Active Comparator 2 — Mango (500 g) + Vitamin C (100 mg)
  Arms: Active Comparator 2
Dietary Supplement: Control Comparator — Vitamin C (100 mg)
  Arms: Control Comparator

SUMMARY:
The primary objectives of the study are:

1. To investigate the relative bioavailability and absorption/kinetic profile of phytochemicals after acute consumption of mango pulp.
2. To study the systemic accumulation or generation of new mango pulp phytochemicals /their metabolites in blood after regular mango intake for an extended time frame.
3. To enhance the bioavailability of polyphenols in mango pulp by addition of Vitamin C to the mango pulp.

DETAILED DESCRIPTION:
The trial is designed as a randomized, 3 arm, within-subject crossover, study design. Subjects meeting eligibility criteria will participate in 3 in-lab visits where they will receive 1 of 3 treatments: Mango (pulp/flesh) (500 g), Mango (500 g) + Vitamin C (100 mg) or Vitamin C (100 mg) only. The study day visit will last for approximately 10.5 h with a follow up visit the next day (24 h) for blood and urine collection to allow for the characterization of target mango pulp phytochemicals and metabolites in plasma and urine. And then after a 2-week wash out period, a 14-day feeding trial will be conducted in which subjects will be given mango pulp (500 g) to take home and instructed to consume every day for 14 days, to study the accumulation of polyphenols and their metabolites in blood. A fasting blood sample will be collected on day 1 of the trial and then again on the 15th day.

Subjects will be required to meet several inclusion and exclusion criteria, which will be assessed through online survey and on-site clinic assessments, including questionnaires, blood analysis and anthropometric measures. Eligible subjects will be invited to participate in the study.

During the Screening Visit, subjects will read, sign and date a written Institutional Review Board approved Informed Consent Form prior to performing any study procedure. And then they will be assessed their qualification, if eligible to participate, subjects will be instructed on the process for completing study questionnaires and counseled to restrict intake of colored plant foods rich in phytonutrients the 7 days prior to each Study Day. They will be asked to restrict alcohol intake, coffee/tea/ caffeinated beverage intake and moderate / vigorous physical activity and to drink plenty of water to maintain hydration in the 24 h prior to each Study Day. They will be instructed to come to the Clinical Nutrition Research Center (CNRC) the day before each Study Day to pick up their dinner meal and evening snack. Subjects will be asked to get a usual night of sleep and to come to the CNRC after a 10-h overnight fasting on each Study Day.

Each study visit will involve with blood samples collection at time points 0 (fasting), 0.5, 1, 2, 3, 4, 6, 7, 8, 9 10 and 24 hour (h) for assessment of change in plasma and metabolites. A drink will be provided immediately after the 0 h blood collection, a breakfast meal will be provided immediately after the 2 h blood collection, and lunch after 6 h blood collection. Urine samples will be collected at 0 (fasting)-2, 2-6, 6-10 and 24 h.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, 20-45 years of age with body mass index (BMI) in range from 20 to 25 kg/m2
* Nonsmokers (Past smokers can be allowed if they have abstinence for minimum of 2 years)
* No clinical evidence of cardiovascular, metabolic, respiratory, renal, gastrointestinal or hepatic disease
* Not taking any medications that would interfere with outcomes of the study, i.e. lipid lowering medications, gastrointestinal medications, antibiotics, anti-inflammatory drugs, dietary supplements including fiber supplements, prebiotics and probiotics, etc.
* Able to provide informed consent
* Able to comply and perform the procedures requested by the protocol (including dietary restrictions, consumption of study treatments, records of food intake and GI-tract questionnaire, sample collection procedures and study visit schedule)

Exclusion Criteria:

* Men and women who smoke
* Men and women with known or suspected intolerance, allergies or hypersensitivity to study foods or treatments
* Men and women known to have/diagnosed with diabetes mellitus
* Men and women who have fasting blood glucose concentrations > 125 mg/dL
* Men and women who have uncontrolled blood pressure >140 mmHg (systolic)/90 mmHg (diastolic)
* Men and women with documented vascular disease, e.g., heart failure, myocardial infarction, stroke, angina, related surgeries, etc. that, in the opinion of the investigator, could interfere with the interpretation of the study results
* Men and women with cancer other than non-melanoma skin cancer in previous 5 years
* Men and women diagnosed with chronic constipation, diarrhea or other chronic gastrointestinal complaint (e.g. irritable bowel syndrome)
* Women who are known to be pregnant or who are intending to become pregnant over the course of the study
* Women who are lactating
* Taking medication or dietary supplements that may interfere with the outcomes of the study; e.g., antioxidant supplement, anti-inflammation, lipid lowering medication, blood pressure lowering medication, etc... Subjects may choose to go off dietary supplements (requires 30 days washout); e.g., fish oil, probiotics, etc...
* Men and women who has participated in prebiotics or laxative trial within 3 months prior to enrollment or any other clinical trial within 1 month
* Men and women who have donated blood within 3 months of the Screening Visit and blood donors/participants for whom participation in this study will result in having donated more than 1500 milliliters of blood in the previous 12 months.
* Men and women who are vegans or vegetarian
* History of an eating disorder (e.g., anorexia nervosa, bulimia nervosa, or binge eating) diagnosed by a health professional
* Substance (alcohol or drug) abuse within the last 2 years
* Excessive coffee and tea consumers (> 5 cups/day)
* Currently eat > 2 servings per day of mangoes
* Men and women who do excessive exercise regularly or athlete
* Unstable weight: gained or lost weight +/- 5 kg (11 lbs) in previous 2 months
* Women who are taking unstable dose and brand of hormonal contraceptives and/or stable dose and brand less than 6 months
* Unusual working hours i.e., working overnight (e.g. 3rd shift)

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2019-05-22 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Characterization of polyphenolic compounds in plasma over 24 h in humans | 24 hr Postprandial
  This will be conducted by using ultra-high performance liquid chromatography iFunnel quadrupole time of flight mass spectrometer (UHPLC-QTOF-MS) and triple quadrupole mass spectrometer (UHPLC-QQQ-MS).

SECONDARY OUTCOMES:
Characterization of Vitamin C in plasma over 24 h in humans | 24 hr Postprandial
  This will be conducted by using ultra-high performance liquid chromatography iFunnel quadrupole time of flight mass spectrometer (UHPLC-QTOF-MS) and triple quadrupole mass spectrometer (UHPLC-QQQ-MS).
Characterization of beta carotene in plasma over 24 h in humans | 24 hr Postprandial
  This will be conducted by using ultra-high performance liquid chromatography iFunnel quadrupole time of flight mass spectrometer (UHPLC-QTOF-MS) and triple quadrupole mass spectrometer (UHPLC-QQQ-MS).
the changes in the metabolite pool following chronic ingestion (14 days) of mango pulp | Baseline vs 2 weeks
  Metabolites will be identified
the bioavailability (Cmax) of polyphenols in mango pulp by addition of Vitamin C to the mango pulp using Cmax. | 24 hr Postprandial
  Cmax will calculated
the bioavailability (AUC) of polyphenols in mango pulp by addition of Vitamin C to the mango pulp using AUC. | 24 hr Postprandial
  Area Under the Curve will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Britt Burton-Freeman, Ph.D, Principal Investigator — Illinois Institute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No